CLINICAL TRIAL: NCT03483311
Title: Estimation of Tissue Level of Resolvin D1 in Psoriasis Before and After Narrowband UVB Phototherapy: a Case-control Study.
Brief Title: Resolvin D1 in Psoriasis Before and After Narrowband UVB Phototherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Fathy Elmasry, principal investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Dermatology7
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- psoriasis patients (Experimental): Tissue levels of resolvin D1 in psoriatic patients before and after NB-UVB.
  Interventions: Other: skin biopsy before and after NB-UVB phototherapy
- controls (Experimental): Tissue levels of resolvin D1 in controls
  Interventions: Other: skin biopsy before and after NB-UVB phototherapy

INTERVENTIONS:
Other: skin biopsy before and after NB-UVB phototherapy — skin biopsy before and after NB-UVB phototherapy to measure tissue resolvin D1

SUMMARY:
• Assessment of tissue level of resolvin D1 in psoriasis in comparison to its level in healthy controls in order to verify its role in the pathogenesis of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with psoriasis (adults and children above 12years)
* Both sexes.
* New cases or cases not receiving any treatment for at least 3 months ago.

Exclusion Criteria:

* Any contraindication to phototherapy treatment (e.g. Photosensitizing creams or medications, past skin cancer, especially melanoma, etc...)
* Erythrodermic and pustular psoriasis.
* History of autoimmune diseases or other systemic diseases (e.g. Alzheimer's disease, fibromyalgia, cystic fibrosis)

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Tissue levels of resolvin D1 in psoriatic patients before and after NB-UVB. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Maha Elmasry, Principal Investigator — Cairo University
Locations (1):
- Maha Fathy Elmasry, Cairo, Egypt

REFERENCES:
- [Derived] Elmasry MF, Hassan E, Rashed LA, Abdel Halim DM. Role of resolvin D1 in psoriasis before and after narrowband ultraviolet B phototherapy: A case-control study. Dermatol Ther. 2021 Mar;34(2):e14879. doi: 10.1111/dth.14879. Epub 2021 Feb 21. PMID 33586174 (Retraction: PMID 34184384 Dermatol Ther. 2021 Jul;34(4):e15038)